CLINICAL TRIAL: NCT01889628
Title: Ethnic Differences in the Glycaemic Response and Glycaemic Index to Liquid-based Nutritional Formulas Between Chinese, Malays and Indians in Singapore
Brief Title: Study to Determine Ethnic Differences in the Glycaemic Response to Nutritional Formula Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Melvin Leow, Associate Professor, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/00403
Record Dates: First submitted 2013-06-21; First posted 2013-06-28 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes; Impaired Glucose Tolerence
Keywords: Glycaemic response; Glycaemic Index; Nutritional formula; Asia; Ethnic differences; Chinese; Malay; Indian
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chinese ethnicity (Other): Three nutritional formulae (Isocal, Protinex and Diasip) and liquid glucose
  Interventions: Dietary Supplement: Liquid-based Nutritional Formulae and liquid glucose
- Malay ethnicity (Other): Three liquid nutritional formulae (Isocal, Diasip and Protinex) and liquid glucose
  Interventions: Dietary Supplement: Liquid-based Nutritional Formulae and liquid glucose
- Indian Ethnicity (Other): Three liquid nutritional formulae (Isocal, Diasip and Protinex) and liquid glucose
  Interventions: Dietary Supplement: Liquid-based Nutritional Formulae and liquid glucose

INTERVENTIONS:
Dietary Supplement: Liquid-based Nutritional Formulae and liquid glucose
  Other Names: Diasip; Protinex; Isocal; liquid glucose

SUMMARY:
Nutritional formula drinks are widely consumed in Asia especially by those having chronic illnesses such as diabetes. Therefore, gauging the impact of nutritional formulas on blood glucose levels is very important. Asia is home to three predominant ethnic groups- Chinese, Malay and Indians. It is still unknown if the blood glucose response to nutritional formulas differs between ethnic groups. Therefore the aim of this study is to observe if there are ethnic differences in the blood glucose response to nutritional formula drinks.

DETAILED DESCRIPTION:
Nutritional formulas are commonly consumed by individuals both to supplement their food intake and as total meal replacers. Consumption rates of nutritional formulas are increasing also in Asia. Very little is known about differences in the glycaemic response to nutritional formulas between different ethnic groups. The aim of the current study is to determine the glycaemic response (GR) and glycaemic index (GI) to three nutrition formulas in Chinese, Indian and Malay subjects.

The study will have a randomised, non-blind, between-subjects, crossover design. The subjects will return for six test sessions. At three random sessions subjects will test the reference food and on the remaining three sessions they will consume the test foods (Diasip, Isocal, Protinex). The first test session will be a glucose test session (for subjects requiring glucose tests). The reference food will be anhydrous glucose (50 g) dissolved in 250 ml of water. The test foods will be portions of the nutritional formulas containing 50 g of available carbohydrates. Subjects who have previously taken part in GI studies at the CNRC and who have already completed three reference glucose tests will have to complete only the three test food sessions. However, they may be asked to do one, two or all three of the glucose tests if their previous test results are old (> 3 months) or are not within the required precision (CV <30%). This aspect will be at the discretion of the investigator and communicated to the participant at the time of briefing (before consenting).

The primary measurement in the study will be the glycaemic response. This will be measured using finger-prick blood samples. The fingers in the non-dominant hand will be used. To encourage blood flow the hand will be warmed using warm water or a hot towel beforehand if required. The finger will then be disinfected using a sterile wipe. Blood will be obtained by finger prick using a single-use lancing device. To minimise plasma dilution fingertips will not be squeezed to extract blood but gently massaged starting from the base of the hand moving towards the tips. The first two drops of expressed blood will be discarded and the next drop (5 μL) will be used for testing. Blood glucose in the sample will be measured using the HemoCue® 201+ Glucose analyser (HemoCue Ltd, Dronfield, UK).

The participants will arrive at the laboratory between 8:30-9 am following a 10 hour overnight fast. They will be instructed not to partake in intense level sports and avoid alcohol consumption on the evening prior to a test session. Following a 10 minute rest two blood samples will be obtained five minutes apart for determining baseline blood glucose levels. If the two baseline blood glucose values are far apart a further 1-2 blood samples may be taken until two stable values are obtained. The study session will be terminated if stable values cannot be obtained or if baseline blood glucose levels are above 6 mmol/L. After obtaining acceptable baseline blood glucose values they will be given either the standard or test food to consume. They will be asked to consume the drink at a comfortable pace within 10 minutes. Further blood samples will be obtained at 15, 30, 45, 60, 90, 120, 150 and 180 minutes for blood glucose measurements. Mandatory sampling will be carried out up to 120 minutes. If the blood glucose level has not reached baseline levels by the end of 120 minutes further samples may be taken at 150 and 180 minutes. During the entire testing period the participants will be instructed to remain rested and in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21-40 years
* Be of Chinese, Malay or Indian ethnic origin
* Do not partake in sports at the competitive and/or endurance levels
* Body mass index between 18 to 24 kg/m2
* Normal blood pressure range (120/80 mmHg)

Exclusion Criteria:

* Those having a fasting blood glucose concentration above 6.0 mmol/l
* Those having metabolic or chronic diseases (Diabetes, hypertension etc)
* Having allergies/intolerances to the foods provided in the study
* Smoking
* Those having medical conditions and/or taking medications known to affect glycaemia or major effects on body fat distribution (glucocorticoids, thyroid hormones, thiazide diuretics)
* Those having gastrointestinal diseases that may interfere with digestion or nutrient absorption
* Those who had medical or surgical events requiring hospitalization within the preceding three months

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Glycaemic response | 2-3 hours post-consumption
  The blood glucose response to the nutritional formula drinks measured over 2-3 hours following their consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Leow, MBBS, Principal Investigator — Institute for Human Development and Potential (IHDP), Singapore
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore, Singapore